CLINICAL TRIAL: NCT05918432
Title: Neuroblastoma Clinical Trials: Looking at Patterns About How Patients Feel About Participating in Clinical Trials
Brief Title: Determining Patterns In Study Experiences of Neuroblastoma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81920705
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in clinical research is highly skewed towards particular demographic groups of people.

This study will invite several participants to gather a wide range of information on clinical trial experiences for neuroblastoma patients. The aim of the study is to identify the factors that limit the ability of a person to enroll in, as well as complete a clinical trial for treatment of neuroblastoma.

The data collected from this study will help improve future outcomes for all neuroblastoma patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of neuroblastoma
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Any serious and/or unstable pre-existing medical disorders
* Enrolled in another research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuroblastoma who are actively considering enrolling in an interventional clinical trial for said condition, but have not yet completed enrollment and randomization phases in said clinical trial.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a neuroblastoma clinical trial | 3 months
Rate of patients who remain in neuroblastoma clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park JR, Kreissman SG, London WB, Naranjo A, Cohn SL, Hogarty MD, Tenney SC, Haas-Kogan D, Shaw PJ, Kraveka JM, Roberts SS, Geiger JD, Doski JJ, Voss SD, Maris JM, Grupp SA, Diller L. Effect of Tandem Autologous Stem Cell Transplant vs Single Transplant on Event-Free Survival in Patients With High-Risk Neuroblastoma: A Randomized Clinical Trial. JAMA. 2019 Aug 27;322(8):746-755. doi: 10.1001/jama.2019.11642. PMID 31454045
- [Background] Park JR, Villablanca JG, Hero B, Kushner BH, Wheatley K, Beiske KH, Ladenstein RL, Baruchel S, Macy ME, Moreno L, Seibel NL, Pearson AD, Matthay KK, Valteau-Couanet D. Early-phase clinical trial eligibility and response evaluation criteria for refractory, relapsed, or progressive neuroblastoma: A consensus statement from the National Cancer Institute Clinical Trials Planning Meeting. Cancer. 2022 Nov 1;128(21):3775-3783. doi: 10.1002/cncr.34445. Epub 2022 Sep 13. PMID 36101004
- [Background] Khomenko VI, Stoliarchuk NP, Ilyk OP. [Reserves of quality]. Veterinariia. 1979 Mar;(3):14-6. No abstract available. Russian. PMID 442501

DOCUMENTS (1):
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT05918432/ICF_000.pdf